CLINICAL TRIAL: NCT05963451
Title: Assessing the Predictability of Brain, Psychological and Epigenetic Determinants for Optimizing the Treatment of Chronic Low Back Pain
Brief Title: Brain, Psychological and Epigenetic Determinants for Optimizing the Treatment of Chronic Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-4293
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva samples to perform epigenetic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Low Back Pain (CLBP) group: Participants who will took part in our study are people living with CLBP who will undergo facet thermal ablation treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be given in our study since, the investigators are recruiting people who will receive already a facet thermal ablation.

SUMMARY:
The goal of this observational study is to better understand the role of the brain in chronic low back pain patients.

DETAILED DESCRIPTION:
Chronic pain affects millions of people worldwide, and the main cardinal sign of any arthritis condition is pain. Several arthritis conditions can cause chronic low back pain (CLBP).The mechanisms that contribute to CLBP are not yet fully understood, but considering the role of the brain in the context of chronic pain, it is only logical to investigate structural and functional brain properties in CLBP, in order to improve diagnosis and treatment of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain (≥ 6 months) with or without pain radiating to the legs or radiating to the neck
* Positive medial branch blocks, suggesting that the pain originates from the lumbar facet joints
* Average pain intensity of ≥ 3/10 in the 24-hour period before the initial visit
* Pain primarily localized in the lower back

Exclusion Criteria:

* Inadequate pain relief or relief of less than three months following selective thermoablation of medial lumbar branches by radiofrequency
* Neurological, cardiovascular, or pulmonary disorders
* Comorbid pain syndrome
* History of surgical intervention in the back
* A corticosteroid infiltration within the past year
* Pregnancy (current or planned during the course of the study)
* Contra-indication to Magnetic Resonance Imaging (MRI)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: -People with CLBP who will have a thermoablation of medial lumbar branches by radiofrequency
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-07 (Estimated); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
Change of Grey matter volume | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  Grey matter volume (milliliters cube) will be measured by acquiring a T1weighted (T1w) image using Magnetic Resonance Imaging.
Change of Blood-oxygen level dependent (BOLD) response | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  Blood-oxygen level dependent (BOLD) response will be measured by using functional Magnetic Resonance Imaging (fMRI).
Change of Microstructural and connectivity properties of white matter tracts | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  Microstructural and connectivity properties will be measured by using diffusion Magnetic Resonance Imaging (dMRI).
Change of Brain's arteries system | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  Brain vasculature will be measured by using Time-of-Flight Magnetic Resonance Angiography (ToF MRA).
Change of Brain's venous system | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  Brain vasculature will be measured by using Susceptibility Weighted Imaging (SWI).

SECONDARY OUTCOMES:
Change of Pain Severity score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Brief Pain Inventory-short form (BPI-SF). Measured on a numerical rating scale (0 = "no pain" to 10 = "worst pain imaginable"). Higher score means worse outcome.
Change of Pain Interference score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Brief Pain Inventory-short form (BPI-SF). Measured on a numerical rating scale (0 = "no interference" to 10 = "complete interference"). Higher score means worse outcome.
Change of Pain Catastrophizing score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Pain Catastrophizing-short form (PCS-SF). Measured on a 5-point Likert-scale (0 = "not at all" to 4 = "all the time"). Higher score means worse outcome.
Change of Neuropathic pain components score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Pain detect. Seven items are measured on a rated on a 6-point Likert Scale (0 = "not at all" to 5 = "very strongly"). Higher score means worse outcome. 1 item based on pain behavior pattern score (-1, 0 or 1) and 1 item based on a radiation score (0 or 2).
Change of Global function score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Pain Outcomes Questionnaire (POQ). Measured on a numeric rating scale (0 = "less symptoms" to 10= "more severe symptoms"). Higher score means worse outcome.
Change of Anxiety score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the State-Trait Anxiety Inventory (STAI-S/T). Measured on a 4-point Likert-scale (0 = "not at all" to 3 = "all the time").
Change of Depression score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Beck Depression Inventory (BDI). Measured on a 4-point Likert-scale (0 = "less symptoms" to 3 = "more severe symptoms"). Higher score means worse outcome.
Change of Fear of movement score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Tampa Scale of Kinesiophobia - short form (TSK-SF).Measured on a 4-point Likert-scale (0 = "Strongly Disagree" to 3 = "Strongly Agree"). Higher score means worse outcome.
Change of Functional disability score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Oswestry Disability Index (ODI). Measured on a 6-point Likert Scale (0 = "less symptoms" to 5 = "more severe symptoms"). Higher score means worse outcome.
Change of Insomnia severity score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Insomnia severity Index (ISI). Measured on a 5-point Likert scale (0 = "not at all" to 4 = "extremely"). Higher score means worse outcome.
Number of traumatic events | Change from Baseline (4 weeks before their treatment) and after their treatment (at 4 months post treatment)
  The investigators will use the Life Events Checklist (LEC). We will count the number of traumatic events.
Patient Expectations score | This will be acquired 1 week before their treatment
  The investigators will use the EXPECT Questionnaire. Measured on numerical rating scale (0 = "no change" to 10 = "complete relief"). Higher score means better outcome.
Change of Global Impression score | Change from Baseline (at 2 months post treatment) and after 2 months (at 4 months post treatment)
  The investigators will use the Patients' Global Impression of Change (PGIC) scale. Measured on numerical rating scale (0 = "no change" to 10 = "complete relief"). Higher score means better outcome.
Change Central sensitization component score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use the Central Sensitization Inventory - short form (CSI-SF). Measured on a 5-point Likert-scale (0 = "never" to 4 = "always"). Higher score means worse outcome.
Patient Gender score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will use a Short Gender Questionnaire (SGQ). Measured on a 5-point Likert-scale (1 = "not at all" to 5 = "extremely").
Change Polygenic methylation score | Change from Baseline (1 week, 2 months and 4 months before their treatment) and after their treatment (at 2 months and 4 months post treatment)
  The investigators will acquire a saliva sample using a DNA kit to perform epigenetic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche du Centre Hospitalier Universitaire de Sherbrooke (CRCHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No